CLINICAL TRIAL: NCT03907163
Title: The Effect of Tetrahydrocannabinol on Ocular Hemodynamics in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: OPHT-141117
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Retinal Blood Flow
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy subjects (Experimental)
  Interventions: Drug: Dronabinol
- healthy volunteers (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dronabinol — Capsules containing 5 mg Dronabinol
  Arms: healthy subjects
Other: Placebo — capsules identical in appearance to dronabinol
  Arms: healthy volunteers

SUMMARY:
Glaucoma is among the leading causes for irreversible blindness worldwide. While lowering intraocular pressure (IOP) remains the mainstay of therapy, there are still some patients who progress despite wellcontrolled IOP. There is evidence from several studies that ocular blood flow and its regulation is impaired in patients with glaucoma. Tetrahydrocannabinol (THC) has been used in the treatment for glaucoma in some countries for several years due to its IOP lowering effect. In addition, there is also evidence that THC features neuroprotective effects and improves ocular hemodynamics. Dronabinol is a synthetic THC that is legally available in several European countries. It has the advantage that exact dosing of THC is possible in contrast to previously applied administration forms such as smoking. Due to its legal status in the past, data about the effect of THC on ocular blood flow and its regulation are sparse. This holds true for basic research in healthy subjects as well as in patients with glaucoma.The aim of the present study therefore is to investigate whether single administration of THC alters optic nerve head (ONH) blood flow in healthy subjects. In addition, other parameters for ocular blood flow will be measured, in particular retinal blood flow, retinal oxygen saturation and retinal neurovascular coupling. The study will be conducted in a randomized, double-masked, placebocontrolled, two-way cross-over design. Subjects will receive 5mg dronabinol on one study day. This dose is the recommended starting dose for some indications in clinical practice. Other studies investigating retinal hemodynamics or IOP after administration of THC also have used similar or slightly higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Normal ophthalmic findings
* Ametropia ≤ 6 diopters
* Normal findings in the medical history and physical examination including ECG unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the laboratory testing unless the investigator considers an abnormality to be clinically irrelevant
* Nonsmokers

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages or drugs
* History of drug or alcohol abuse
* Psychiatric disorders in the medical history
* Risk for drug dependence as evaluated by a psychiatrist
* Participation in a clinical trial in the 3 weeks preceding the study
* Positive urine drug test at the screening examination or on the study days
* Positive alcohol breath test at the screening examination or on the study days
* Regular consumption of cannabis and inability to not consume cannabis during the study period
* Treatment in the previous 3 weeks with any drug (except intake of oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Known hypersensitivity to any of the components of the IMP under investigation or other study medication
* History or family history of epilepsy
* Pregnant or breast-feeding women
* Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (oral contraceptives, intra-uterine device, contraceptive implant or condoms)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow | 60 minutes
  To determine the total blood flow in the eye, OCT measurements were performed with a rectangular scanning pattern around the optical nerve head.

OTHER OUTCOMES:
Retinal vessel diameter (DVA) | 30 minutes
  The DVA allows for the real time measurement of retinal vessel diameters in vivo.
  The DVA is a commercially available system (IMEDOS, Jena, Germany) which comprises a fundus camera, a video camera, a real time monitor and a personal computer with an analyzing software for the accurate determination of retinal arterial and venous diameters. Every second a maximum of 25 readings of vessel diameter can be obtained. For this purpose the fundus is imaged onto the charge coupled device chip of the video camera. The consecutive fundus images are digitized using a frame grabber. In addition, the fundus image can be inspected on the real time monitor and, if necessary, stored on a video recorder. Evaluation of the retinal vessel diameters can either be done online or offline from the recorded video tapes
Retinal oxygen saturation (DVA) | 30 minutes
  In particular, retinal oxygen saturation measurement is based on the image analysis by the DVA software of two monochromatic fundus images as recorded by a standard DVA. In an image, obtained by the camera and filter assembly, the operator has to mark the vessel of interest by a mouse click. The vessel is traced automatically applying the following procedure. The vessel walls are located as photometric edges in the vicinity of the mouse cursor in the green channel image. If edges are determined, the search is continued in their proximity.
Retinal blood velocities | 15 minutes
  We observe bi-directional blood flow and pulsatility of blood velocity in retinal vessels with a Doppler detection bandwidth of 12.5 kHz and a longitudinal velocity sensitivity in tissue of 200μm/s.
THC plasma concentration | 120 minutes
  Measurements of ocular hemodynamics will be started one hour after administration, since maximum plasma levels are reached 60-120 minutes after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University Vienna, Vienna, Austria